CLINICAL TRIAL: NCT05110690
Title: Behavioral Activation and Medication Optimization for Perioperative Mental Health Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101103; 1P50MH122351 (NIH)
Record Dates: First submitted 2021-10-18; First posted 2021-11-08 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Older Adults; Anxiety; Depression; Cardiac Surgery; Orthopedic Surgery; Major Surgical Resection of a Thoracic Malignancy; Major Surgical Resection of an Abdominal Malignancy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Participants (Experimental): * Behavioral activation (BA) will span across 3 months postoperatively & will begin pre-operatively, with sessions approximately weekly or biweekly, depending on patient preference & health condition.
  * Medications will be reviewed & optimized by a team of interventionists including a psychiatrist, pharmacologist, & pharmacists. While the participant is in-hospital, the interventionist's role will include coordinating with the hospital team to ensure that medication changes that were introduced preoperatively are maintained in-house & that no new inappropriate medications are initiated. After discharge, & up to approximately 3 months postoperatively, the interventionist will ensure that medication changes are reconciled during transitions of care. The interventionists will ensure the agreed-upon changes are implemented, or an alternative course of action is justified.
  Interventions: Behavioral: Behavioral Activation; Other: Medication Optimization

INTERVENTIONS:
Behavioral: Behavioral Activation — The behavioral intervention will consist of behavioral activation (BA), the basic premise of which is to help people with mental health problems to engage in activities that are reinforcing or meaningful and guided by their personal values
Other: Medication Optimization — Medication optimization consists of a simple set of principles: reconcile patient's medications, identify the patient's likely need for, and interest in, a medication adjustment, make the adjustment, and assess the response to that adjustment.

SUMMARY:
Inadequate management of preoperative mental health disorders often contributes to poor postoperative outcomes, including increased rates of readmission, delirium, falls, and mortality. However, very little work has been done to improve perioperative mental health. In particular, there have been limited systematic efforts that identify evidence-based behavioral and pharmacological strategies that were originally developed for depression and anxiety in otherwise medically well psychiatric patients. A mental health intervention bundle, composed of behavioral and pharmacological strategies, can mitigate anxiety and depression symptoms during the perioperative period. However, lacking is conclusive evidence on effectiveness of such an intervention bundle focused on the delivery of perioperative mental health care in older surgical patients. Towards this end, the investigators will develop and test an intervention bundle that encompasses: (1) behavioral activation, and (2) medication optimization.

DETAILED DESCRIPTION:
The proposed research is relevant to public health because the prevalence of undertreated depression/anxiety in older adults coupled with the increasing number of surgeries performed in this population are creating a crucial need for the integration of mental health interventions into critical periods, such as the perioperative period. Thus, the proposed research is relevant to the mission of the NIMH to transform the treatment of mental illnesses through clinical research, paving the way for prevention, recovery, and cure.

ELIGIBILITY:
Inclusion Criteria Patient Participants

* Age ≥60 years on the day of surgery;
* Scheduled major orthopedic surgery, or major surgical resection of a thoracic or abdominal malignancy, or major cardiac procedure;
* Clinically significant depression or anxiety symptoms screened by the PHQ-ADS (Patient Health Questionnaire Anxiety and Depression Scale) ≥10

Exclusion Criteria Patient Participants

* Estimated life expectancy < 12 months;
* Unable to read, speak, and understand English;
* Current alcohol or other substance abuse;
* Severe cognitive impairment screened by the SBT (Short Blessed Test) >10;
* Acutely suicidal

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Avidan, MBBCh, FCASA, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abraham J, Meng A, Baumann A, Holzer KJ, Lenard E, Freedland KE, Lenze EJ, Avidan MS, Politi MC. A multi- and mixed-method adaptation study of a patient-centered perioperative mental health intervention bundle. BMC Health Serv Res. 2023 Oct 27;23(1):1175. doi: 10.1186/s12913-023-10186-3. PMID 37891574
- [Derived] Abraham J, Holzer KJ, Lenard EM, Freedland KE, Tellor Pennington BR, Wolfe RC, Cordner TA, Baumann AA, Politi M, Avidan MS, Lenze E. Perioperative mental health intervention bundle for older surgical patients: protocol for an intervention development and feasibility study. BMJ Open. 2022 Aug 23;12(8):e062398. doi: 10.1136/bmjopen-2022-062398. PMID 35998971
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the primary outcome measure, the number of participants eligible for consent and enrollment (n=29 participants) needs to be indicated in the participant flow.
Period: Eligible for Consent and Enrollment
Arm/Group | Patient Participants
Started | 29
Completed | 24
Not Completed | 5
Not completed — Did not consent | 5
Period: Enrolled
Arm/Group | Patient Participants
Started | 24
Completed | 24
Not Completed | 0
Period: Started Intervention
Arm/Group | Patient Participants
Started | 24
Completed | 23
Not Completed | 1
Not completed — Ineligible due to canceled surgery | 1
Period: Completion of Intervention
Arm/Group | Patient Participants
Started | 23
Completed | 19
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patient Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Reach of the Study as Measured by the Number of Participants Who Agree to Participate in the Study Out of the Total Eligible Participants
Time Frame: Through completion of the study (13 months and 5 days)
Population: One participant who signed consent, was considered eligible, and was enrolled to the study ended up having their surgery canceled and became ineligible for the study after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 28
Participants | 23

2. Primary Outcome: Reach of the Intervention Bundle as Measured by the Number of Participants Who Completed the Intervention Out of the Participants Who Agreed to Participate in the Study
Time Frame: Through completion of the study (13 months and 5 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 23
Participants | 19

3. Secondary Outcome: Completeness of Planned Primary Outcome Data Collection at Specified Timepoints as Measured by the Number of Participants Who Completed 100% of the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS)
Time Frame: Baseline, 1 month, and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 23
Participants
  Baseline | 23
  1 month | 15
  3 months | 20

ADVERSE EVENTS:
Time Frame: From start of intervention through completion of intervention (up to 3 months).
Arm/Group | Patient Participants
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05110690/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT05110690/ICF_001.pdf